CLINICAL TRIAL: NCT01942031
Title: An Interventional Study of How Collegial Feed Back to Primary Care Physicians on Detection of Diagnosis and Dispensation of Prescribed Secondary Preventive Drugs Affect Stroke Prevention.
Brief Title: Improved Prevention of Stroke in Primary Care in Stockholm, Sweden (Förbättrad Prevention av Stroke)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mia von Euler, Associate Professor, Head Karolinska Institutet Stroke Research Network at Södersjukhuset, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPN2010/1158-31/2
Record Dates: First submitted 2013-04-15; First posted 2013-09-13 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke; TIA; Atrial Fibrillation
Keywords: Ischemic stroke; Hemorrhagic stroke; TIA; Atrial fibrillation; prevention; primary care
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- structured collegial feed back (Experimental): Structured feed back and information about stroke to the primary care center, to physicians and head of the center
  Interventions: Behavioral: structured collegial feed back
- Control group (No Intervention): No structured feed back on stroke prevention. Ordinary educational activities only.

INTERVENTIONS:
Behavioral: structured collegial feed back — Collegial feed back to primary care physicians at randomized primary care centers
  Arms: structured collegial feed back

SUMMARY:
Stroke is a devastating disease. The acute mortality in Sweden is 20 % and 25 % of all patients relapse. Secondary prevention is proven efficient but observational studies have shown that a number of patients are lost to follow up and do not receive recommended prevention. The aim of the study is to 1) describe, by analyzing register data, the detection rate of patients with hospital diagnosis of stroke, TIA, and atrial fibrillation in the primary care center where they are listed. The analysis is done by sex, age, and socioeconomic status. Furthermore, rate of dispensed prescriptions of secondary preventive drugs are analysed for the identified population. 2) in a randomized controlled study evaluate if collegial feed back and targeted information of secondary prevention to the intervention group can improve the detection rate and the medication of the patients listed at the participating primary care centers.

DETAILED DESCRIPTION:
All primary care centers in Stockholm County (approximately 200) are randomised to control or intervention (receiving structured feed back on detection rate of stroke/transient ischemic attacks in comparison to hospital discharge registry data. The randomisation is done group wise based on training areas. A data set is presented by different means; 1) in written reports, directly to the head of each primary care center in the intervention group 2)in oral presentation on training sessions for the physicians in each training ares. Measures of detection rates of diagnosis and dispensed prescriptions of secondary preventive drugs are made before start of the project and after one year. The control group, ie the primary care centers not receiving feed back, are measured in the same way and thus provide a control group. The hypothesis being that with visibility of the problem, it is easier to improve care wich is what all health providers aim to do.

Outcome measures is percentage of patients with stroke (ICD code I60, I 61, I63, I64) and transitory ischemic attacks(G45) who are dispensed prescribed secondary preventive medication and death.

ELIGIBILITY:
Inclusion Criteria:

* Primary care center in Stockholm county

Exclusion Criteria:

* localisation outside Stockholm County

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-10; Primary Completion 2019-03 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
percentage of identified patients with stroke/TIA in primary care and analysis of dispensed prescriptions in each group | Outcome meassures will be followed during two years
  percentage of patients identified with hospital discharge diagnosis of stroke/TIA in primary care diagnosis register. Analysis of changes in outcome before intervention and after. the intervention will take place during one year and collection of data before start of intervention and one year after ended intervention will be performed

SECONDARY OUTCOMES:
dispensed prescriptions of secondary preventives drugs in patients with stroke/TIA | baseline 2010 and 2012, followed for one year after intervention
  dispensed prescriptions of recommended secondary preventive drugs in patients detected and not detected at each primary care center

CONTACTS AND LOCATIONS:
Overall Officials: Mia von Euler, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Stroke Research Network at Södersjukhuset, Stockholm, Sweden

REFERENCES:
- [Result] Geary L, Hasselstrom J, Carlsson AC, Eriksson I, von Euler M. Secondary prevention after stroke/transient ischemic attack: A randomized audit and feedback trial. Acta Neurol Scand. 2019 Aug;140(2):107-115. doi: 10.1111/ane.13109. Epub 2019 May 9. PMID 31017305
- [Result] Geary L, Hasselstrom J, Carlsson AC, Schenck-Gustafsson K, von Euler M. An audit & feedback intervention for improved anticoagulant use in patients with atrial fibrillation in primary care. Int J Cardiol. 2020 Jul 1;310:67-72. doi: 10.1016/j.ijcard.2020.04.027. Epub 2020 Apr 12. No abstract available. PMID 32327203